CLINICAL TRIAL: NCT07061119
Title: Effect of Cawthorne Cooksey Exercises on Balance in Autistic Children With Vestibular Hypofunction.
Acronym: ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bushra Zahid
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Vestibular Hypofunction
Keywords: Autism, vestibular rehab in children, Autism and balance
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Interventional model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Conventional treatment include: Trampoline jumping Gym ball exercise:5reps'Sensory diet: Joint compressions Deeppressure Balance board exercises
  Interventions: Other: Conventional treatment
- Participant Group (Experimental): Cawthorne cooksey exercises
  Interventions: Other: cawthorne cooksey exercises

INTERVENTIONS:
Other: Conventional treatment — Trampolinejumping:5times. Gym ball exercise:5reps'Sensory diet:- Joint compressions: 1 set x 10reps on limbs, neck, and head region.
  Deeppressure:1 setx10reps. Balance board exercises.
  Arms: Conventional treatment
Other: cawthorne cooksey exercises — Cawthorne Cooksey exercises
  * Start with low to moderate intensity.
  * Gradually increase range, speed, and Complexity over time
  * Trampoline jumping- Gym ball exercise- Sensory diet
  * Cawthorne Cooksey exer cise Training
  Phase1-In bed exerercises:- Eye movements:
  1)Up and down 2)Side to side 3)Moving finger away from face
  * Phase2-Sitting: Eye movements as above. Head movements at firsts low, then quick later with eyes closed
  * bending forward and backward
  * turning from side to side.
    --Shoulder shrugging and circling
  * Bending forward and picking up objects from the ground
  * Phase 3 - Standing:
  * Eye, Head, Shoulder movements
  * Throwing ball from hand to hand, hand under knee
  * Switch to sitting to standing and turning around in between.
  * Phase 4 - Walk: with eyes closed and open:
  * Across room
  * Slope and Stairs
  Arms: Participant Group

SUMMARY:
The objective of the study is to determine the effects of cawthorne cooksey exercises on balance in autistic children with vestibular hypofunction. The study will be randomized control trial including 2 experimental groups with estimated 22 participants in each group.

DETAILED DESCRIPTION:
The complex neurodevelopmental disorder known as autism spectrum disorder (ASD) affects people in a variety of ways, affecting their ability for social interaction, communication, and repetitive behavior. Typically, ASD is recognized and diagnosed in the early childhood years, although its impact can extend throughout a person's life. Autism Spectrum Disorder (ASD) is a type of condition that affects how a child's brain develops. It appears that they have a somewhat different brain than others, which may have an impact on their behavior, social interactions, and communication. It can involve repetitive actions and a strong focus on specific interests. Symptoms of autism differ from person to person depending on age and ability that's why it is called spectrum disorder. Children with autism spectrum disorder appear to exhibit altered postural control when facing challenging situations. Postural control predominantly relies on the automatic system, necessitates focused attention during various straightforward or intricate tasks, and facilitates the regulation of postural control.

Vestibular functioning refers to operation and effectiveness of vestibular system, which is normally concerned with spatial orientation, movement, and balance. The system is located in the inner ear and comprises of semicircular canals (fluid-filled canals) and sensory receptors. Vestibular dysfunction is another common manifestation is autistic patients. It refers to impaired ability to sense and process sensory information associated with balance, movement, and spatial orientation. The manifestations of vestibular dysfunction include apprehensive behaviors when feet do not touch the ground, avoidance of jumping/climbing, and escaping activities like playing with playground equipment. The children usually exhibit toe walking and take more risks while playing. Interventions to improve balance due to vestibular dysfunction include trampoline Jumping, Gym ball exercises, balance board exercises. Balance issues play a huge role in life of an individual with autism. There is indeed a huge gap and lack of literature on how or if exercise protocols from physical therapy can influence balance in individuals with autism. Although, Previous studies have recommended that Balance issues and autism are directly related and that vestibular dysfunction plays a huge role in maintenance of posture. The aim of the study is to investigate the effects of Cawthorne Cooksey exercises on balance. This study will also influence how a physical therapist can improve quality of life of an individual with autism by improving their balance

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Peripheral Vestibular hypofunction.
* Age:7-15years
* Children with mild to moderate autism.
* Children who understand and communicate

Exclusion Criteria:

* Central Vestibular.
* Acute Infection of inner ear
* Auditory issues.
* Patients unable to follow exercise plan

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | 6 Weeks
  Adapted from the Berg Balance Scale for pediatric use.Assesses flexibility in changing postures and overall postures. - Comprises 14 different balance- related tasks, scored from 0 to 4. Used to assess functional balance skills and motor disorders in school-aged children.
CTSIB-M | 6 Weeks
  This test is aimed to asses' sensory input when one or more sensory system is compromised. It Assess balance (either vestibular or non- vestibular). It consists of 4 different conditions; 4 conditions e.g. eye open/ eye close and firm surface. Eyes open/ eye close foam surface. each consist of 3 trials. Total time 30 sec for each trial and total score is 120. Excellent reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS, Principal Investigator — Riphah International University
Locations (1):
- Islamabad, Pakistan, Islamabad, Fedral, Pakistan

REFERENCES:
- [Background] Lord C, Brugha TS, Charman T, Cusack J, Dumas G, Frazier T, Jones EJH, Jones RM, Pickles A, State MW, Taylor JL, Veenstra-VanderWeele J. Autism spectrum disorder. Nat Rev Dis Primers. 2020 Jan 16;6(1):5. doi: 10.1038/s41572-019-0138-4. PMID 31949163
- [Background] Mughal S, Faizy RM, Saadabadi A. Autism spectrum disorder. 2018